CLINICAL TRIAL: NCT06281587
Title: Pathogenetic Risk Factors for Corneal Graft Rejection in Penetrating Keratoplasty Patients
Brief Title: Pathogenetic Risk Factors for Corneal Graft Rejection
Status: Completed | Type: Observational
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Responsible Party: Principal Investigator, Alexander Romanov, Head of the Department, The S.N. Fyodorov Eye Microsurgery State Institution
Other Study IDs: SNFyodorov
Record Dates: First submitted 2024-01-31; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Graft Rejection
Keywords: penetrating keratoplasty; corneal graft rejection; corneal opacity; risk factors
MeSH Terms: conditions — Corneal Opacity | interventions — Keratoplasty, Penetrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - low-risk (LR) keratoplasty: if the patient was diagnosed with keratoconus and there were no concomitant complicating diagnoses (n = 42)
  Interventions: Procedure: penetrating keratoplasty
- Group 2 - high-risk (HR) keratoplasty: in the presence of corneal dystrophy (pseudophakic bullous keratopathy, primary dystrophy), corneal inflammatory pathology (erosions, corneal ulcers, corneal fistulas,leucoma), complicated keratoconus, CGR or rekeratoplasty (n = 51)
  Interventions: Procedure: penetrating keratoplasty

INTERVENTIONS:
Procedure: penetrating keratoplasty — replacement of the affected tissue with healthy donor tissue in diseases that disrupt the shape or transparency of the cornea.

SUMMARY:
There are many predictors that may influence the development of corneal graft rejection after penetrating keratoplasty. In our study investigators analysed the results of keratoplasty and the risk factors for graft rejection.

Investigators analysed data from 493 patients who underwent penetrating keratoplasty between 2011 and 2019. Keratoplasty outcomes were followed up at subsequent clinic visits until December 2021. Then, 93 medical records were selected (taking into account the completeness of the medical records) and divided into two groups based on the primary diagnosis that was an indication for keratoplasty: high-risk and low-risk patients. Investigators then estimated the survival time (clear graft) of the corneal graft using Kaplan-Meier statistical survival analysis. Investigators also investigated the factors that influence corneal graft opacity.

DETAILED DESCRIPTION:
The pathogenesis of corneal graft rejection (CGR) is complex and is associated with numerous risk factors related to the donor, recipient and surgical technique.

Donor-related factors. These include AB0 and HLA incompatibility. Compared to corneal transplantation from a male donor to a male recipient, corneal transplantation from a male donor to a female recipient is associated with HR (high risk) CGR. Factors such as the method of storage of the donor cornea, sex mismatch between recipient and donor, and cause of death of the donor are not thought to have a significant impact on the outcome of keratoplasty. However, storage of donor tissue in organ culture medium for 7 days or more may reduce the incidence CGR.

Recipient-related factors. The most important risk factor for corneal graft rejection is the degree of corneal neovascularization (CNV) in the recipient. Another risk factor is rekeratoplasty. The presence of chronic diseases - herpes keratitis, uveitis, atopic dermatitis - also increases the risk of immune reactions. Dry eye syndrome (DES) and a history of glaucoma increase the risk of keratoplasty rejection. The presence of antibodies after rejection of other previously transplanted organs and blood transfusions can significantly increase the risk of rejection. Low limbal stem cell counts due to degradation of the limbal palisades of Vogt may lead to poor re-epithelialisation and development of corneal damage in the post-operative period.

Surgical factors. It has been observed that penetrating keratoplasty (PKP) has a lower graft survival rate than lamellar keratoplasty (LKP).

The aim of this study was to analyse the results of keratoplasty and to identify the risk factors for post-operative opacities of the corneal graft.

The study was conducted in accordance with the ethical standards of the authors' institutions and the Declaration of Helsinki (revised in 2013) and was approved by the Local Biomedical Ethics Committee of the The S.N. Fyodorov Eye Microsurgery State Institution no. 1 from 11.09.2019. Written informed consent was not required for participation in the study. The study was retrospective and patient data were anonymised.

Study design and groups The data of patients (n = 493) with corneal surgeries performed in " ISTC "Eye Microsurgery" named after Acad. S.N. Fedorov" Krasnodar for the period from 2011 to 2019. The results of keratoplasty were tracked at the patients' subsequent visits to the clinic until December 2021. Thus, the study included data from 8 years of postoperative follow-up of the patients.

In the next step, 93 medical records were selected from the entire cohort of patients who underwent penetrating keratoplasty (PKP), taking into account the completeness of data and records. These cases were divided into two groups without randomisation according to the primary diagnosis that indicated keratoplasty:

* Group 1 - low-risk (LR) keratoplasty - if the patient was diagnosed with keratoconus and there were no concomitant complicating diagnoses (n = 42);
* Group 2 - high-risk (HR) keratoplasty - in the presence of corneal dystrophy (pseudophakic bullous keratopathy, primary dystrophy), corneal inflammatory pathology (erosions, corneal ulcers, corneal fistulas,leucoma), complicated keratoconus, CGR or rekeratoplasty (n = 51).

Pharmacological management postoperative Antibiotics, antiseptics, keratoprotectors and Lubricating Eye Drops and gels were used for postoperative pharmacological management.

Methods of clinical evaluation of keratoplasty outcomes In the overall cohort group, recipient-related factors (ophthalmological and somatic status), primary and concomitant diagnoses, type of keratoplasty and postoperative complications were assessed.

In the next step, diagnostic data of the patients' ophthalmological examinations were obtained from electronic medical records and archives: examination and consultation by an ophthalmologist, refractometry, keratometry, visometry, tonometry, endothelial cell density (ECD), Schirmer test, optical coherence tomography (OCT) of the anterior segment, as well as graft characteristics and incidence of postoperative complications.

In groups 1 and 2, the assessment of graft transparency at each visit and signs of CGR, if present, were recorded in the medical records. CGR (or postoperative graft opacity) was defined if rekeratoplasty was performed and the loss of central graft transparency caused visual impairment for at least three consecutive months, if the patient's database or medical record mentioned the development of CGR as a diagnosis or postoperative complication. Stages of data analysis: 0 - at hospital admission before keratoplasty, 1, 3, 6, 9, 12 months after surgery. The anatomical results of keratoplasty (clear graft or postoperative graft opacity) in the cohort group and in groups 1 LR and 2 HR - were evaluated during the follow-up period of 8 years.

ELIGIBILITY:
Inclusion Criteria:

* completeness of data and records

Exclusion Criteria:

* no

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: corneal inflammatory pathology (erosions, corneal ulcers, corneal fistulas,leucoma), complicated keratoconus, CGR or rekeratoplasty
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Cohort group Kaplan-Meier survival analysis (clear graft engraftment) | 2011-2019
  Investigators used Kaplan-Meier survival analysis to evaluate the survival (clear graft) of the corneal graft in this cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Krasnodar, Russia

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make the iPad available.

REFERENCES:
- [Result] Inoue K, Tsuru T. ABO antigen blood-group compatibility and allograft rejection in corneal transplantation. Acta Ophthalmol Scand. 1999 Oct;77(5):495-9. doi: 10.1034/j.1600-0420.1999.770501.x. PMID 10551286
- [Result] Di Zazzo A, Kheirkhah A, Abud TB, Goyal S, Dana R. Management of high-risk corneal transplantation. Surv Ophthalmol. 2017 Nov-Dec;62(6):816-827. doi: 10.1016/j.survophthal.2016.12.010. Epub 2016 Dec 22. PMID 28012874
- [Result] Guilbert E, Laroche L, Borderie V. [Rejection of corneal allografts]. J Fr Ophtalmol. 2011 May;34(5):331-48. doi: 10.1016/j.jfo.2011.02.001. Epub 2011 Apr 14. French. PMID 21492957
- [Result] Hopkinson CL, Romano V, Kaye RA, Steger B, Stewart RM, Tsagkataki M, Jones MN, Larkin DF, Kaye SB; National Health Service Blood Transplant Ocular Tissue Advisory Group and Contributing Ophthalmologists (OTAG Study 20). The Influence of Donor and Recipient Gender Incompatibility on Corneal Transplant Rejection and Failure. Am J Transplant. 2017 Jan;17(1):210-217. doi: 10.1111/ajt.13926. Epub 2016 Jul 22. PMID 27412098
- [Result] Simon M, Fellner P, El-Shabrawi Y, Ardjomand N. Influence of donor storage time on corneal allograft survival. Ophthalmology. 2004 Aug;111(8):1534-8. doi: 10.1016/j.ophtha.2003.12.060. PMID 15288984
- [Result] Writing Committee for the Cornea Donor Study Research Group; Sugar A, Gal RL, Kollman C, Raghinaru D, Dontchev M, Croasdale CR, Feder RS, Holland EJ, Lass JH, Macy JI, Mannis MJ, Smith PW, Soukiasian SH, Beck RW. Factors associated with corneal graft survival in the cornea donor study. JAMA Ophthalmol. 2015 Mar;133(3):246-54. doi: 10.1001/jamaophthalmol.2014.3923. PMID 25322173
- [Result] Armitage WJ, Goodchild C, Griffin MD, Gunn DJ, Hjortdal J, Lohan P, Murphy CC, Pleyer U, Ritter T, Tole DM, Vabres B. High-risk Corneal Transplantation: Recent Developments and Future Possibilities. Transplantation. 2019 Dec;103(12):2468-2478. doi: 10.1097/TP.0000000000002938. PMID 31765363
- [Result] Yamaguchi T, Higa K, Tsubota K, Shimazaki J. Elevation of preoperative recipient aqueous cytokine levels in eyes with primary graft failure after corneal transplantation. Mol Vis. 2018 Sep 13;24:613-620. eCollection 2018. PMID 30262982
- [Result] Siebelmann S, Ramos SL, Matthaei M, Scholz P, Schrittenlocher S, Heindl LM, Bachmann B, Cursiefen C. Factors Associated With Early Graft Detachment in Primary Descemet Membrane Endothelial Keratoplasty. Am J Ophthalmol. 2018 Aug;192:249-250. doi: 10.1016/j.ajo.2018.05.010. Epub 2018 May 29. No abstract available. PMID 29858043